CLINICAL TRIAL: NCT04683354
Title: A Phase I, Open-Label, Multi-Center Dose Escalation Study to Evaluate Safety, Pharmacokinetics and Preliminary Efficacy of HL-085 in Patients With Advanced Solid Tumors
Brief Title: Study of HL-085 in Patients With Advanced Solid Tumor Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kechow Pharma, Inc. (Industry)
Responsible Party: Sponsor
Organization: Shanghai Kechow Pharma, Inc. (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HL-085-US-102
Record Dates: First submitted 2020-11-30; First posted 2020-12-24 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental): There are 3 cohorts for the dose escalation study. Six subjects each cohort will receive oral administration of HL-085 capsules at three daily dose levels (12 mg, 18 mg and 24 mg). Three subjects of each cohort will receive TID and 3 subjects will receive BID dose regimen. Dose escalation can occur after 6 patients have completed 28 days of treatment and no or 1 DLT is identified.
  Interventions: Drug: HL-085

INTERVENTIONS:
Drug: HL-085 — HL-085 is a MEK inhibitor with potential indication for cancers. It will be given twice or three times daily continuously in the study until disease progression; or the risks outweigh the benefits, if the subject continues study treatment; or subjects with poor compliance; or subjects need to receive or have already started alternative antitumor drugs; or Subjects who need to receive or have already started alternative any other concomitant medication and/or treatment, which would significantly impact their safety; or interruption of IP administration for more than 14 days due to IP-related AEs.

SUMMARY:
The investigational product (IP) HL-085 is an adenosine triphosphate-noncompetitive mitogen activated protein kinase (MEK) inhibitor with a strong selective anti-tumor activity, with a much lower dose than selumetinib. It has been shown strong anti-tumor activities in preclinical studies to treat solid tumors, e.g., melanoma, non-small cell lung cancer, colon cancer and other malignancies with RAF and RAS mutations.

Kechow has completed phase I dose escalation study to test HL-085 in patients with advanced NRAS mutated melanoma in China. The tested doses were 0.5 mg, 1mg, 2mg, 3mg, 4mg, 6mg, 9mg, 12mg, 15mg and 18mg BID oral administration and there was no dose-limiting toxicity (DLT) identified. All patients tolerated the study drug reasonably well.

This study is a Phase I, open-label, dose escalation study to evaluate tolerability, safety, pharmacokinetic (PK) and preliminary antitumor activities of HL-085 in US patients with advanced solid tumors. The objective of the dose escalation is to evaluate safety and tolerability of selected TID and BID dose regimens in US patient population with advanced solid tumor and establish the Recommended Phase 2 Dose (RP2D).

The starting dose for this trial is 12 mg daily oral administration. Three selected daily doses - 12 mg (4mg TID, 6mg BID), 18 mg (6mg TID, 9 mg BID), and 24 mg (8 mg TID, 12 mg BID) will be tested in this study to assess safety and tolerability of HL-085 at the 3 selected dose levels in US patient population with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained prior to any clinical trial procedures
2. Aged 18 years or over.
3. Must have a pathologically documented solid tumor(s) that has relapsed from, or is refractory to standard treatment, or unable to tolerate toxicities from the SOC/available treatments, or for which no standard treatment is available.
4. Must have at least one measurable lesion as defined by RECISTv1.1 criteria for solid tumors.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
6. Life expectancy ≥3 months (as judged by the Investigator).
7. Must have adequate hematologic function (no blood transfusion and growth factor support for ≥14 days), adequate hepatic and renal function, and some key lab test results meeting the following laboratory values within 7 (+/-2) days before first dosing.
8. Must have the willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedures.

Exclusion Criteria:

1. Have biological, chemotherapy, immunotherapy or radiotherapy less than 4 weeks prior to starting the study treatment.
2. Have undergone or plan to have major surgery (except for tumor biopsy) or experienced severe trauma ≤28 days prior to starting the study treatment.
3. Have active central nervous system lesion (i.e., imaging instability and neurologically unstable). Note: patients who have received stereotactic radiotherapy or surgical treatment for brain tumor can be included after 3 months of procedure without symptoms.
4. Previous or history of second malignancy within 3 years prior to study treatment except for curatively treated.
5. Prior therapy with MEK-inhibitor with severe toxicity causing permanent damage from it, such as ocular, cardiac, pulmonary, etc. disorders and illness.
6. History of any of the following within 6 months prior to Screening:

   * Myocardial infarction.
   * Unstable angina.
   * Coronary artery bypass graft.
   * Coronary angioplasty or stenting.
   * Chronic heart failure (New York Heart Association Grade ≥2).
   * Ventricular arrhythmias requiring continuous therapy.
   * Supraventricular arrhythmias, including atrial fibrillation, which are uncontrolled.
   * Uncontrolled hypertension despite optimal medication management (per Investigator's assessment)
   * Cerebrovascular accidents including transient ischemic attack, or pulmonary embolism.
   * Creatine Phosphokinase (CPK) >2.5×ULN due to underlying cardiac disorders or myocardial infarction.
7. Mean resting QT calculated using Bazzetts formula (QTcB) ≥480 obtained from three electrocardiograms (ECGs); or family or personal history of long or short QT syndrome; Brugada syndrome or known history of QTc prolongation or Torsade de Pointes within 12 months of Screening.
8. Left ventricular ejection fraction (LVEF) <50%.
9. History or current evidence of retinal diseases (e.g., retinal vein occlusion [RVO] or retinal pigment epithelial detachment, macular degeneration, and retinal detachment).
10. Active/chronic infection with hepatitis C (note: patients positive for anti hepatitis C virus [HCV] antibody will be eligible if they are negative for HCV-ribonucleic acid [HCV-RNA]); or active hepatitis B, or active/chronic infection with human immunodeficiency virus (HIV).
11. Known active tuberculosis.
12. Infectious diseases requiring systemic treatment including patients tested positive for COVID-19 according to investigator site/institution's COVID-19 management policies and guidelines.
13. History of allogeneic bone marrow transplantation or organ transplantation.
14. Interstitial lung disease or interstitial pneumonitis, including clinically significant radiation pneumonitis (i.e., affecting activities of daily living or requiring therapeutic intervention). Patients with subclinical pneumonitis who have received immunotherapy previously can be included if his/her condition is stable without any medical intervention.
15. Known hypersensitivity to IP ingredients or their analogues.
16. Unable to swallow IP or has refractory nausea and vomiting, malabsorption, external biliary diversion, or any significant small bowel resection that may interfere with adequate absorption of IP.
17. Concomitant medication which are strong inducers or strong inhibitors of cytochrome P450 CYP2C9, CYP2C19, CYP 3A4.
18. Pregnant or breast-feeding females.
19. Female patients of child-bearing potential or male patients who will not use an effective form of contraception for the duration of the study (until at least 30 days after the last dose of study medication).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Characterize the safety profile of the study drug at 3 dose levels in terms of number of treatment emergent events assessed by CTCAE v5.0., abnormal clinical laboratory and electrocardiograms findings (i.e. QT and QTc intervals). | 7 months (6 months treatment + 1 month follow-up)
Cmax: the maximum plasma concentration of HL-085 or metabolite(s); | 1 month (Cycle 1 Day 1-31)
Tmax: the time of Cmax; | 1 month (Cycle 1 Day 1-31)
Area under the curve at steady state: a measure of the exposure to HL-085 or metabolite(s) at steady state. | 1 month (Cycle 1 Day 1-31)

SECONDARY OUTCOMES:
Evaluate the efficacy of the study drug in terms of overall response rate, progression-free survival. ORR is the proportion of patients with a best overall response of complete response (CR) or partial response (PR), as assessed per RECIST v1.1. | 7 months (6 months treatment + 1 month follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Hongqi Tian, PhD, Study Director — Kechow Pharma, Inc.
Locations (5):
- United States (5):
  - CCARE, San Marcos, California
  - Comprehensive Cancer Centers, Las Vegas, Nevada
  - Gabrail Cancer Center, Canton, Ohio
  - SCRI, Nashville, Tennessee
  - Oncology Consultants, Houston, Texas

IPD SHARING:
Plan to Share IPD: No